CLINICAL TRIAL: NCT06338124
Title: Value of Laboratory Biomarkers in Prediction of Outcome in Septic Patients
Status: Recruiting | Type: Observational
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Other Study IDs: David Ibrahim
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- survivor group: About 50 patients whom will be relifed from the sepsis and will be discharged from the Intensive Care Unit
  Interventions: Diagnostic Test: Triglyceride glucose index
- non-survivor group: About 50 patients whom will be died from the sepsis in the Intensive Care Unit
  Interventions: Diagnostic Test: Triglyceride glucose index

INTERVENTIONS:
Diagnostic Test: Triglyceride glucose index — To evaluate the role of various laboratory biomarkers ( TyG , RAR , CAR, N\L ratio, CRP, Serum lactate )in prediction of sepsis outcome.

SUMMARY:
Sepsis is defined as a dysregulated host response to infection . Despite ongoing efforts, both the incidence and mortality of sepsis have demonstrated limited reductions over the past years,There are several biomarkers that have already been studied for the early diagnosis of sepsis. Some of these markers can be used in risk prediction and monitoring the outcome of sepsis .

Some of these markers as procalcitonin and CD14, are costly and not feasible options for low- and middle-income countries . While other biomarkers are feasible and accessible to be evaluated as Triglyceride\glucose index (TyG) , Relative Distributive Width of red blood corpuscles to albumin ratio (RAR), C-reactive protein,Neutrophile \Lympocyte ratio and serum lactate levels .

DETAILED DESCRIPTION:
Sepsis is defined as a dysregulated host response to infection . Despite ongoing efforts, both the incidence and mortality of sepsis have demonstrated limited reductions over the past years,

There are several biomarkers that have already been studied for the early diagnosis of sepsis. Some of these markers can be used in risk prediction and monitoring the outcome of sepsis .

Triglyceride-glucose (TyG) index has emerged as a surrogate marker of insulin resistance which is often prevalent in patients with sepsis. Red blood cell distribution width (RDW) is a common clinical hematology indicator that reflects the heterogeneity of red blood cell size. As a simple and inexpensive parameter, RDW has been successfully used to predict the prognosis of many diseases, including cardiovascular disease, kidney disease, diabetes mellitus, and liver disease .

Recent studies have also shown that RDW is significantly associated with the mortality of sepsis. RDW to albumin ratio was evaluated as a novel and simple biomarker of inflammation.

-C-reactive protein (CRP) is a sensitive indicator of the body, reflecting damage and infection .

Serum albumin level drops significantly in the acute stage of infection (16). CRP/ALB ratio (CAR) could be a marker to predict mortality in sepsis.

The neutrophil-lymphocyte ratio (NLR) is an-inflammatory biomarker that can be used as an indicator of systemic inflammation. It is a simple that does not add costs to complete blood count laboratory examinations, which are performed routinely in hospitals. It was tested as a guide for the prognosis of various diseases, such as cancer, community pneumonia and sepsis.

Although these various biomarkers that have been proposed, no single clinical or biological indicator of sepsis has gained general acceptance . And to our knowledge, no previous study compared between these indicators in prediction of sepsis outcome or determined the clinical significance of combination of multiple biomarkers in prognosis of sepsis .

ELIGIBILITY:
Inclusion Criteria:

- patients whom will be diagnosed with sepsis

Exclusion Criteria:

* patients diagnosed by hematological disease
* patients refused to participate in the research
* patients less than 18 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To evaluate the role of various laboratory biomarkers ( TyG , RAR , CAR, N\L ratio, CRP, Serum lactate )in prediction of sepsis outcome
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Mortality Outcome Measure | 28 days
  Number of Participants whom will be diagnosed with sepsis and will be admitted in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Fatema Abu-Bakre, Professor, Study Chair — Internal medicine, faculty of medicine, Assuit University,Egypt
Locations (1):
- Assuit University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided